CLINICAL TRIAL: NCT05622461
Title: Setting Families on a Positive Path to Recovery After Pediatric TBI: Road-to-Recovery, A Randomized Control Trial
Brief Title: Setting Families on a Positive Path to Recovery After Pediatric TBI: Road-to-Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0221
Record Dates: First submitted 2022-10-24; First posted 2022-11-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury; Head Injury; Head Injuries, Closed; Brain Hemorrhage, Traumatic; Brain Edema; Intracranial Edema
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Head Injuries, Closed; Brain Hemorrhage, Traumatic; Brain Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Road-to-recovery group (R2R) (Experimental): Usual medical care plus the R2R-TBI intervention (self-guided web-program)
  Interventions: Behavioral: Road-to-recovery
- Internet resources comparison group (IRC) (Active Comparator): Usual medical care plus internet resources
  Interventions: Behavioral: Road-to-recovery

INTERVENTIONS:
Behavioral: Road-to-recovery — R2R-TBI is a self-guided web-based intervention that targets caregiver psychological functioning, parenting behaviors, and family functioning in the first three months following pediatric traumatic brain injury.

SUMMARY:
This study has two main goals: 1) to refine and enhance the R2R-TBI intervention; and 2) to examine the efficacy of the R2R-TBI intervention in a randomized control trial. To achieve the second goal, we will employ a between-groups randomized treatment design with repeated measures at baseline, one-month post-randomization, and at a six-month follow-up. The two conditions will be: a) usual medical care plus access to internet resources regarding pediatric brain injury (Internet Resources Comparison group, IRC), and b) usual medical care plus the R2R-TBI intervention (Road-to-Recovery group, R2R-TBI).

DETAILED DESCRIPTION:
The early recovery period constitutes a critical window to set families on a positive road-to-recovery by supporting parental self-care, positive parent-child interactions, and awareness of potential longer-term concerns. The latter would facilitate parental recognition of behavioral and psychosocial needs that might otherwise go unmet.

Recognizing that (1) caregivers of children who have sustained TBI are at risk of worsening psychological health and that (2) caregiver functioning and parenting behaviors have a direct impact on child recovery and outcomes; intervening and supporting caregivers in the acute phase following injury may set children and families on a positive path to recovery. Intervening at the acute phase may reduce the cascading effects of parental burden/distress and concomitant negative parent-child interactions on child recovery and functioning over time.

Because families of children with TBI and other chronic health conditions may have difficulty accessing services due to transportation and cost issues, particularly lower income families, the R2R-TBI program is designed to be accessed via any web-enabled device (e.g., smartphone, computer, tablet) with any form of internet connection. We will also offer the intervention (via tablet) to parents while they wait for their child to complete outpatient therapies (e.g., speech, physical, and occupational therapy). Delivery of web-based behavioral health interventions may reduce barriers to help-seeking and promote evidence-based interventions that are both accessible and efficient.

ELIGIBILITY:
Inclusion Criteria:

Caregivers will be eligible if they are over 18 years of age, and if their child meets all of the following criteria:

* Ages 3 months to 18 years at time of discharge from hospital
* Sustained a complicated mild to severe TBI as defined by a Glasgow Coma Scale (GCS) of 13-15 with imagining abnormalities or GCS 3-12 with or without imaging abnormalities
* Admitted overnight to the hospital
* 0-3 months post-discharge

Exclusion Criteria:

The caregiver will be excluded from participation if any of the following occur:

* Child did not survive the injury
* Child sustained a non-blunt head trauma (e.g. gunshot wound)
* Child does not reside with parent/caregiver for study duration
* English is not primary language spoken in the home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Parent anxiety | Change from baseline at 4-6 weeks post-intervention
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Measure 4a; scores range from 4-20 with higher score indicating greater symptoms of anxiety
Parent anxiety | Change from baseline at 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Measure 4a; scores range from 4-20 with higher score indicating greater symptoms of anxiety
Parent depression | Change from baseline at 4-6 weeks post-intervention
  Center for Epidemiological Studies Depression Scale (CES-D; 10-items); scores range from 0 -30 with higher scores indicating of higher levels of depressive symptomatology
Parent depression | Change from baseline at 6 months
  Center for Epidemiological Studies Depression Scale (CES-D; 10-items); scores range from 0 -30 with higher scores indicating of higher levels of depressive symptomatology
Parenting self-efficacy | Change from baseline at 4-6 weeks post-intervention
  Caregiver self-efficacy scale (CSES); scores range from 25-100, higher scores indicate greater parenting self efficacy
Parenting self-efficacy | Change from baseline at 6 months
  Caregiver self-efficacy scale (CSES); scores range from 25-100, higher scores indicate greater parenting self efficacy
Parent post-traumatic symptoms | Change from baseline at 4-6 weeks post-intervention
  Primary Care PTSD Screen for DSM-5 (PC-PTSD-5); scores rage from 0-5 with higher scores indicating greater experience of post-traumatic stress symptoms
Parent post-traumatic symptoms | Change from baseline at 6 months
  Primary Care PTSD Screen for DSM-5 (PC-PTSD-5); scores rage from 0-5 with higher scores indicating greater experience of post-traumatic stress symptoms

SECONDARY OUTCOMES:
Family Functioning | Change from baseline at 4-6 weeks post-intervention
  Family Assessment Device - Global Functioning Scale. Scores range from 1 to 4 with higher scores indicating poorer family functioning
Family Functioning | Change from baseline at 6 months
  Family Assessment Device - Global Functioning Scale. Scores range from 1 to 4 with higher scores indicating poorer family functioning
Family Burden of Injury | Change from baseline at 4-6 weeks post-intervention
  Family Burden of Injury Interview (FBII). Average scores range from 0-4; higher scores indicate greater injury-related burden
Family Burden of Injury | Change from baseline at 6 months
  Family Burden of Injury Interview (FBII). Average scores range from 0-4; higher scores indicate greater injury-related burden
Child Socioemotional Functioning | Change from baseline at 4-6 weeks post-intervention
  Pediatric Quality of Life Scale (PEDS-QL) - Psychosocial Health Summary Score (score range varies based on child age; higher scores indicate greater health related quality of life)
Child Socioemotional Functioning | Change from baseline at 6 months
  Pediatric Quality of Life Scale (PEDS-QL) - Psychosocial Health Summary Score (score range varies based on child age; higher scores indicate greater health related quality of life)
Parent mindful self-care | Change from baseline at 4-6 weeks post-intervention
  Mindful self-care scale (MSCS); scores range from 6 - 30, higher scores denote greater frequency in engaging in self-care behaviors
Parent mindful self-care | Change from baseline at 6 months
  Mindful self-care scale (MSCS); scores range from 6 - 30, higher scores denote greater frequency in engaging in self-care behaviors
Parent resilience | Change from baseline at 4-6 weeks post-intervention
  Connor-Davidson Resilience Scale (CDRI); scores range from 0-40 with higher scored indicating greater resilience
Parent resilience | Change from baseline at 6 months
  Connor-Davidson Resilience Scale (CDRI); scores range from 0-40 with higher scored indicating greater resilience

OTHER OUTCOMES:
Moderators of treatment effects | 4-6 weeks
  Examining household income and baseline caregiver distress as moderator of treatment effects
Moderators of treatment effects | 6 months
  Examining household income and baseline caregiver distress as moderator of treatment effects

CONTACTS AND LOCATIONS:
Overall Officials: Shari Wade, PhD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share deidentified data as consistent with requirement of funding source (i.e., The National Institute on Disability and Rehabilitation Research).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: Plan is to share deidentified data as consistent with protocols of funding source (i.e., The National Institute on Disability and Rehabilitation Research).